CLINICAL TRIAL: NCT05410847
Title: A Prospective Study of Intraperitoneal and Intravenous Nab-paclitaxel Plus Camrelizumab and S-1 Conversion Therapy for Gastric Cancer With Positive Exfoliative Cancer Cells
Brief Title: Nab-paclitaxel Plus Camrelizumab and S-1 Conversion Therapy for Gastric Cancer With Positive Exfoliative Cancer Cells
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Hebei Medical University (Other)
Responsible Party: Principal Investigator, Qun Zhao, Principal Investigator, Hebei Medical University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: HRCG-001
Record Dates: First submitted 2022-06-06; First posted 2022-06-08 (Actual); Last update posted 2022-06-24 (Actual); Status verified 2022-06

CONDITIONS: Gastric Cancer
MeSH Terms: conditions — Stomach Neoplasms

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Experimental (Experimental): Camrelizumab: 200mg，iv，30min, q3w, 4 cycles. Nab-Paclitaxel: intraperitoneal nab-paclitaxel 80 mg/m2 and intravenous nab-paclitaxel 180 mg/m2 on days 1, q3w, 4 cycles.
  S-1：According to the body surface area, BSA <1.25m2，40mg bid; 1.25m2≤BSA≤1.5m2，50mg bid; BSA >1.5m2, 60mg bid. Take the medicine twice daily for 2 weeks, then suspend for 1 week, q3w, 4 cycles.
  For patients who were operable, the original regimen was continued for 4 cycles of adjuvant treatment after operation, followed by maintenance of carrelizumab monotherapy to 1 year.
  Inoperable patients were selected for follow-up treatment according to guidelines recommended by the investigator.
  Interventions: Drug: Camrelizumab Nab-Paclitaxel S-1

INTERVENTIONS:
Drug: Camrelizumab Nab-Paclitaxel S-1 — Camrelizumab+S-1+Intraperitoneal nab-paclitaxel and intravenous nab-paclitaxel

SUMMARY:
The purpose of this study is to investigate the efficacy and safety of intraperitoneal and intravenous nab-paclitaxel plus Camrelizumab and S-1 conversion therapy for gastric cancer with positive exfoliative cancer cells.

ELIGIBILITY:
Inclusion Criteria:

1. None previous chemotherapy, radiotherapy and other antitumor therapy;
2. Age:18 to 70 years old;
3. Man or female (except pregnant and lactating women);
4. Conﬁrmed to gastric adenocarcinoma and HER2-negative;
5. Proven gastric cancer of T stage was T3 and T4, and no distant metastasis was observed. The exfoliative cancer cells detection in peritoneal washes was positive;
6. Blood cell count has to meet the following certeria:

   WBC≥3.5×109/L; ANC≥1.5×109/L; PLT≥100×109/L; HB≥90g/L;
7. Liver/kidney function has to meet the following certeria:

   ALT and AST≤2.5×ULN TBIL<1.5×ULN； Serum creatinine ≤1.5×ULN;
8. Left ventricular ejection fraction (LVEF) ≥50%;
9. Eastern Cooperative Oncology Group (ECOG) performance status of 0-1;
10. Participants were willing to join in this study, good adherence and written informed consent.

Exclusion Criteria:

1. Subjects with immunosuppressive medications within 14 days of first administration of study treatment, excluding nasal spray and inhaled corticosteroids or physiological doses of systemic steroid hormones (no more than 10 mg / day of prednisolone or other corticosteroids of equivalent pharmaceutical physiological dose);
2. The patient has any active autoimmune disease or a history of autoimmune disease (such as the following, but not limited to: autoimmune hepatitis, interstitial pneumonia, uveitis, enteritis, hepatitis, pituitary inflammation, vasculitis, nephritis, hyperthyroidism, hypothyroidism; patients with vitiligo; Asthma has been completely relieved in childhood, and patients who do not need any intervention after adulthood can be included; asthma patients who require bronchodilators for medical intervention cannot be included);
3. Patients with other malignant tumors within 5 years;
4. Human immunodeficiency virus (HIV) infection or acquired immunodeficiency syndrome (AIDS), active hepatitis B (HBV-DNA ≥1000 IU/ml) or hepatitis C (positive hepatitis C antibody, and HCV-RNA is higher than the lower limit of detection of the analytical method) or co-infection with hepatitis B and C, requiring antiviral treatment during the study;
5. Distant metastasis;
6. It has serious or uncontrolled medical diseases and infections (Including atrial fibrillation, angina pectoris, cardiac insufficiency, ejection fraction less than 50%, poor-controlled hypertension and so on);
7. History of psychiatric drugs abuse and can't quit or patients with mental disorders;
8. Patients with severe or uncontrollable mental illness;
9. It have serious harm to the patient's safety or affect the patients who have completed the research.
10. The researchers think inappropriate.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2022-06-30 (Estimated); Primary Completion 2023-06-30 (Estimated); Study Completion 2025-06-30 (Estimated)

PRIMARY OUTCOMES:
R0-resection rate | within 3 weeks after surgery
  There was no residual by the microscope
Conversion to negative rate | within 3 weeks after surgery
  Exfoliative cytology positive gastric cancer conversion to negative rate

SECONDARY OUTCOMES:
Overall survival (OS) | 3years
  Baseline to measured date of death from any cause
Progression free survival (PFS) | 3years
  Baseline to measured date of progression or death from any cause
Objective response rate (ORR) | tumor assessment every 6 weeks since the treatment began，up to 3years
  Baseline to measured stable disease
Disease control rate (DCR) | tumor assessment every 6 weeks since the treatment began，up to 3years
  Baseline to measured progressive disease
Tumor regression grade (TRG) | within 3 weeks after surgery
  TRG included four grades: Grade 0-3
Adverse events | 3 years
  Toxicity according to the Common Terminology Criteria for Adverse Events (CTCAE) Version 5.0. The number of Participants with adverse events will be recorded at each treatment visit.

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Lv J, Wu J, Wu H, Ding P, Guo H, Yang P, Tian Y, Liu Y, Zhao Q. Study protocol of a phase II clinical trial evaluating the efficacy of neoadjuvant intraperitoneal and systemic albumin-bound paclitaxel combined with camrelizumab and S-1 in the treatment of patients with exfoliative cell-positive gastric cancer. Front Oncol. 2023 Sep 29;13:1201928. doi: 10.3389/fonc.2023.1201928. eCollection 2023. PMID 37841441